CLINICAL TRIAL: NCT04946617
Title: The Effect of Chlorhexidine and Essential Oil Mouthwashes on Human Beta-Defensin 2 (hbD2) and Kathelicidin (LL-37) Saliva Levels
Brief Title: Chlorhexidine and Essential Oil Mouthwashes on Human Beta-Defensin 2 (hbD2) and Kathelicidin (LL-37) Saliva Levels
Acronym: hbD2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mustafa Cihan Yavuz, Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 9.2.2017-30
Record Dates: First submitted 2021-06-14; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Mouth and Tooth Diseases; Periodontal Diseases; Gingivitis
Keywords: Periodontitis; Gingivitis; Mouthwashes
MeSH Terms: conditions — Stomatognathic Diseases; Periodontal Diseases; Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- H group: healthy periodontium, BOP at \20 % of the sites and no sites with probing depth (PD) [3 mm and clinical attachment level (CAL) [2 mm or alveolar bone loss (N = 20, 12 males, 8 females, mean age: 33.38
  Interventions: Drug: undefined
- G group: gingivitis, BOP at ≥20 % of the sites and no sites with PD and CAL [3 mm or bone loss (N = 20, 6 males, 14 females, mean age: 32.35);
  Interventions: Drug: undefined
- CP group: chronic periodontitis, ≥4 teeth in each jaw with PD of ≥5 mm, CAL of C4 mm, BOP at [≥80 % of the proximal sites and radiographic evidence of interproximal bone loss
  Interventions: Drug: undefined

INTERVENTIONS:
Drug: undefined — Rinsing with mouthwashes
  Other Names: Mouthwash Product

SUMMARY:
Recent studies have shown that while mouthwashes exhibit antimicrobial properties against bacteria and their products, at the same time showing the cytotoxic effect on living cells in the mouth.29 To the best of our knowledge, there is no information about the toxicity effect of these two mouthwashes, which are highly preferred, on antimicrobial peptides secreted from the oral epithelium. Therefore, our aim in this study is to evaluate the effect of chlorhexidine and essential oil mouthwash on hBD2 and LL-37 in saliva.

DETAILED DESCRIPTION:
Periodontal health continues with a balanced interaction of the oral microflora with the host defense line.

ELIGIBILITY:
Inclusion Criteria:

1. systemically healthy,
2. presence of ≥20 natural teeth,
3. agreement to participate in the study .

Exclusion Criteria:

1. known systemic illness,
2. smoking habit,
3. pregnancy/ lactation,
4. long-term use of anti-inflammatory drugs.

Ages: 25 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: The sample size was calculated using (power of 80%). The present study included 40 patients per group (total of 120) to have a power >80%.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of periodontal parametres changes | 6 Months
  Incidence of Gingivitis
Rate of periodontal parametres changes | 6 Months
  Incidence of Periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa C Yavuz, PhD, Principal Investigator — Istanbul Medeniyet University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Dyke TE. Pro-resolving mediators in the regulation of periodontal disease. Mol Aspects Med. 2017 Dec;58:21-36. doi: 10.1016/j.mam.2017.04.006. Epub 2017 May 18. PMID 28483532